CLINICAL TRIAL: NCT07213167
Title: Clinical Evaluation of Low Contrast Defocus Curves, Low Light Photic Phenomena, and Dysphotopsia Profiles in Pseudophakic Patients
Brief Title: Clinical Evaluation of Low Contrast Visual Performance and Low Light Phenomena in Patients With Various Intraocular Lens Implants
Status: Recruiting | Type: Observational
Sponsor: Dr. Daniel H. Chang, MD (Other)
Collaborators: Johnson & Johnson Surgical Vision, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Dr. Daniel H. Chang, MD, Principal Investigator, Empire Eye and Laser Center
Organization: Empire Eye and Laser Center (Other)
Other Study IDs: EMP-2025-001
Record Dates: First submitted 2025-09-24; First posted 2025-10-08 (Actual); Last update posted 2025-10-08 (Actual); Status verified 2025-10

CONDITIONS: Dysphotopsia; Posterior Capsule Opacification; Visual Acuity; Visual Function; Contrast Sensitivity
Keywords: Dysphotopsia; Posterior Capsule Opacification; Halometry; Manifold Vision Meter; PRVSQ; AIOLIS; TECNIS Eyhance IOL; TECNIS Symfony Optiblue IOL; TECNIS Odyssey IOL; Low Contrast; Defocus Curves; Low Light Photic Phenomena; Dysphotopsia Profiles; Pseudophakia
MeSH Terms: conditions — Pseudophakia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (3):
- Tecnis Eyhance: Pseudophakic subjects with Tecnis Eyhance, model DIB00, DIUxxx intraocular lenses.
  Interventions: Other: None-placebo
- Tecnis Symfony Optiblue: Pseudophakic subjects with Tecnis Symfony Optiblue, model ZXR00V, ZXWxxx intraocular lenses.
  Interventions: Other: None-placebo
- Tecnis Odyssey: Pseudophakic subjects with Tecnis Odyssey, model DRN00V, DRTxxx intraocular lenses.
  Interventions: Other: None-placebo

INTERVENTIONS:
Other: None-placebo — No interventions.

SUMMARY:
The goal of this clinical investigation is to evaluate visual acuity and contrast sensitivity in low lighting conditions using several different testing devices, and measure nighttime side effects of intraocular lens (IOL) implants after cataract surgery.

Researchers will compare the results for three different types of IOLs to see how each lens contributes to overall visual function, patient experience and satisfaction.

Participants will:

* Complete two different questionnaires about their current vision
* Undergo visual testing using several different devices

DETAILED DESCRIPTION:
The purpose of the study is to correlate the low contrast defocus curves, objective halometry measurement of low light photic phenomena, and patient reported dysphotopsia profiles of the various study IOLs.

The primary endpoints are low (50%) contrast defocus curve, halometry (cool white light) assessment of photic phenomena, and PRVSQv2 results.

The secondary endpoints are:

* Visual Acuity
* BCDVA
* Low contrast (50%) BCDVA
* Contrast Sensitivity
* High contrast defocus curve
* Halometry:
* Light levels: low, medium, high
* Colors: cool white, warm white, red, green
* Characterization of glare, starbursts, and halos
* PRO questionnaires
* AIOLIS
* Patient satisfaction and recommendation survey
* Pupil size
* YAG capsulotomy within 1 year
* Posterior capsular opacification: pre-planned post-hoc analysis evaluating performance in patients w/wo PCO Monocular BCDVA

Participants will:

* Complete PRVSQ v2 and AIOLIS vision questionnaires in a randomized order.
* Undergo the following visual testing using M&S, clinical halometry, and the manifold vision meter devices:
* Manifest refraction
* Distance visual acuity
* Defocus testing
* Low contrast testing
* Contrast sensitivity
* Pupilometry
* Halometry
* Biomicroscopic slit-lamp exam
* Intraocular pressure
* Non-directed ocular symptoms

ELIGIBILITY:
Inclusion Criteria:

* Minimum 22 years of age
* Bilateral pseudophakia, at least 3 months postoperative from IOL implantation, with one of the study IOL models in at least one eye.
* Availability, willingness, and sufficient cognitive awareness to comply with examination procedures
* Signed informed consent and HIPAA authorization or equivalent documentation necessary to comply with applicable privacy laws pertaining to medical treatment in the governing countries
* Ability to understand and respond to a questionnaire in English

Exclusion Criteria:

* Any clinically significant pupil abnormalities (non-reactive, fixed pupils, or abnormally shaped pupils.
* Inability to focus or fixate for prolonged periods of time (e.g., due to strabismus, nystagmus, etc.)
* Uncorrected distance visual acuity worse than 20/25 in either eye
* Prior corneal refractive surgery (LASIK, LASEK, RK, PRK, etc.) or intraocular surgery. Note: Prophylactic peripheral iridotomies and peripheral laser retinal repairs that, in the opinion of the investigator will not confound study outcomes are acceptable.
* Posterior capsular opacification with grading worse than 1+
* Ocular findings that may, in the opinion of the investigator, affect vision and/or contrast sensitivity

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Bilateral pseudophakia, at least 3 months postoperative from IOL implantation with one of the study IOL models.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2025-09-24 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Low (50%) contrast defocus curve | Day 1
  Measured low (50%) contrast defocus curve compared between all three groups
Halometry assessment of photic phenomena | Day 1
  Halometry assessment of halos and starbursts utilizing a cool white light with varying intensities. Comparing the measured size of the ring (deg) of each condition between all three groups.
PRVSQv2 questionnaire results | Day 1
  PRVSQv2 questionnaire results compared between all three groups:
  Frequency and bother/severity of symptoms (scale 1 to 5, with 5 most bothersome)

SECONDARY OUTCOMES:
Best corrected distance visual acuity (BCDVA) | Day 1
  Best corrected distance visual acuity (BCDVA) compared between all three groups
Low contrast (50%) BCDVA | Day 1
  Low contrast (50%) BCDVA compared between all three groups
Contrast Sensitivity | Day 1
  Contrast sensitivity compared between all three groups
High Contrast Defocus Curve | Day 1
  High Contrast Defocus Curve compared between all three groups
Halometry | Day 1
  Halometry assessment of halos and starbursts utilizing various light colors (cool white, warm white, red, yellow, and green) and intensities. Comparing the measured size of the ring (deg) of each condition between all three groups.
Patient-Reported Outcome (PRO) Questionnaires | Day 1
  PRVSQv2 and AIOLIS vision questionnaire results compared between all three groups. Frequency and bother/severity of symptoms (scale 1 to 5, with 5 most bothersome)
Pupil Size | Day 1
  Photopic and mesopic pupil size compared between all three study groups
YAG Capsulotomies | Day 1
  Number of YAG capsulotomies performed within one year post-op compared between all three groups
Posterior capsular opacification (PCO) | Day 1
  Pre-planned post-hoc analysis evaluating number of participants with and without PCO compared between all three groups

CONTACTS AND LOCATIONS:
Overall Officials: Daniel H Chang, MD, Principal Investigator — Empire Eye and Laser Center
Locations (1):
- Empire Eye and Laser Center, Bakersfield, California, United States

IPD SHARING:
Plan to Share IPD: No